CLINICAL TRIAL: NCT03488602
Title: A Focused Suicide Prevention Strategy for Youth Presenting to the Emergency Department With Suicide Related Behaviour: A Randomized Controlled Trial
Brief Title: Focused Suicide Prevention Strategy for Youth
Acronym: FSPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Cundill Centre for Child and Youth Depression (Unknown); SickKids Foundation (Other)
Responsible Party: Principal Investigator, Daphne Korczak, Psychiatrist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000056892
Record Dates: First submitted 2018-02-08; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research staff responsible for measuring outcomes will be blinded to participants' randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-SPS Intervention (Experimental): This group will receive the F-SPS intervention.
  Interventions: Behavioral: F-SPS+UC
- Enhanced Usual Care (EUC) (Active Comparator): This group will receive Enhanced Usual Care (EUC)
  Interventions: Behavioral: EUC

INTERVENTIONS:
Behavioral: F-SPS+UC — Manualized individual and family program. Weekly individual and family sessions with a therapist for 6 weeks.
  Participants will continue to receive usual care.
  Other Names: F-SPS + UC
  Arms: F-SPS Intervention
Behavioral: EUC — Weekly telephone contact with parents regarding participant health care utilization. Referrals to community mental health resources provided as needed.
  Participants will continue to receive usual care.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study evaluates whether a Family-centered suicide prevention strategy, when added to usual care (F-SPS + UC), is more effective than enhanced usual care (EUC) in reducing suicide-related behaviors in 128 youth at high-risk of suicide. Half of the participants will be randomized to receive F-SPS + UC and half will receive EUC.

DETAILED DESCRIPTION:
This is a RCT of a patient- and family-centered suicide prevention intervention added to usual care (F-SPS + UC) for adolescents aged 12 to 18 years who present to the Emergency Department (ED) with suicidal ideation or suicide risk behaviours. The investigators will determine whether the F-SPS + UC intervention is more effective than enhanced usual care (EUC) in reducing suicide-related behaviors in 128 youth at high-risk of suicide.

F-SPS is a 6-week, standardized, manualized outpatient program that teaches participants to the skills to manage suicidal thoughts and impulses effectively. The family component addresses conflictual relationships that may be present in the family as well as improving family communication.

Enhanced usual care consists of 6 weekly telephone calls to ensure that the participant has connected with community resources suggested by the ED team and provide additional resources as needed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to18 years
* Youth presenting in the Emergency Department with acute suicidal ideation or suicide risk behaviour
* SIQ-Jr score ≥ 31
* Parent or caregiver able to communicate in English, or is willing to communicate using a hospital-organized translator, and willing to participate in study
* Living in the greater Toronto area and access to a telephone.

Exclusion Criteria:

* Active psychosis or hypomania/mania
* Moderate to severe intellectual disability, autism.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation severity as measured by the Suicidal Ideation Questionnaire - Jr | Screening, 6 weeks, 24 weeks
  a 15-item measure self-report of suicide ideation (e.g., thoughts about death and dying) completed by the patient. Items are scored from 0 to 6, yielding a score from 0 to 90. Higher scores indicate more severe suicidal ideation.

SECONDARY OUTCOMES:
Change in suicide related behavior as measured by the Suicide Behavior Questionnaire - Revised | Screening, 6 weeks, 24 weeks
  A 4-item self-report questionnaire that measures suicide behavior, and yields a total score of 3 - 18. Higher scores indicate more severe suicidal behavior.
Changes in emotional regulation using the Life Problems Inventory | Baseline, 6 weeks, 24 weeks
  A 60-item self-report scale that measures emotional regulation on a 5 point Likert scale from 1 to 5. Higher scores indicate more impaired emotional regulation. The measure has four subscales: Confusion about Self, Impulsivity, Emotion Dysregulation, and Interpersonal Chaos. Each subscale has a score from 15 to 75 where a higher score indicates more severity.
Change in family conflict as measured by the Conflict Behavior Questionnaire | Baseline, 6 weeks, 24 weeks
  A 20-item scale that examines the parent-child relationship using true/false ratings, yielding a total score of 0 to 20. Higher scores This measure is completed by both the youth and the parent(s) or caregiver. Higher scores indicate more severe family conflict.
Changes in global impairment as measured by the Columbia Impairment Scale | Baseline, 6 weeks, 24 weeks
  A 13-item scale designed to measure functioning on a 5 point Likert scale from 0 to 4, yielding a total score of 0 to 52. This measure is completed by both the youth and the parent(s) or caregiver. Higher scores indicate more severe impairment.
Changes in affect regulation as measured by the Children's Affective Lability Scale | Baseline, 6 weeks, 24 weeks
  A 20-item parent-report instrument that measures difficulties with emotion regulation on 5 point Likert scale from 0 to 4, yielding a score from 0 to 80. Higher scores indicate more severe affective lability.
Health Care Utilization Survey | Baseline, 24 weeks
  A parent-report qualitative interview of a youth's use of available health care services, medication, and the costs associated with those services.
Usual Care Tracking Survey | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
  A parent-report qualitative interview of a youth's use of available health care services over a 1 week period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne J Korczak, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Matthew Tracey, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Tracey M, Finkelstein Y, Schachter R, Cleverley K, Monga S, Barwick M, Szatmari P, Moretti ME, Willan A, Henderson J, Korczak DJ. Recruitment of adolescents with suicidal ideation in the emergency department: lessons from a randomized controlled pilot trial of a youth suicide prevention intervention. BMC Med Res Methodol. 2020 Sep 14;20(1):231. doi: 10.1186/s12874-020-01117-5. PMID 32928140
- [Derived] Korczak DJ, Finkelstein Y, Barwick M, Chaim G, Cleverley K, Henderson J, Monga S, Moretti ME, Willan A, Szatmari P. A suicide prevention strategy for youth presenting to the emergency department with suicide related behaviour: protocol for a randomized controlled trial. BMC Psychiatry. 2020 Jan 14;20(1):20. doi: 10.1186/s12888-019-2422-y. PMID 31937274

DOCUMENTS (2):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT03488602/Prot_000.pdf
  • Informed Consent Form (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT03488602/ICF_001.pdf